CLINICAL TRIAL: NCT03190239
Title: Efficacy and Safety of Maintenance Apatinib Combined With Pemetrexed After First - Line Induction Chemotherapy in Advanced Non-squamous Non-small Cell Lung Cancer: A Prospective, Open, Single Arm Clinical Study
Brief Title: Efficacy and Safety of Maintenance Apatinib Combined With Pemetrexed in Advanced Non-squamous Non-small Cell Lung Cancer Patients
Acronym: XQonc-007
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: abandon
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Professor, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-007
Record Dates: First submitted 2017-05-12; First posted 2017-06-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Advanced Non-squamous Non-small-cell Lung Cancer
MeSH Terms: interventions — apatinib; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib XQonc-0007 (Experimental): Pemetrexed 500 mg/m2, qm; Apatinib 250 mg Po qd
  Interventions: Drug: Apatinib; Drug: Pemetrexed

INTERVENTIONS:
Drug: Apatinib — Apatinib 250mg qd
Drug: Pemetrexed — Pemetrexed 500mg/m2 qm

SUMMARY:
Lung cancer is a malignant tumor that causes the highest morbidity and mortality, and the main pathological type is non-small cell lung cancer (NSCLC). Most of them present with advanced stage at diagnosis. This design is to study maintenance therapy with pemetrexed plus apatinib after first line induction therapy four cycles for advanced non-squamous non-small-cell lung cancer. XQonc-0007

DETAILED DESCRIPTION:
XQonc-0007

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologic confirmed，locally advanced and/or metastatic non-squamous NSCLC of stage IIIB or IV or recurrent NSCLC
2. At least one measurable lesion
3. If genetic testing (EGFR/ALK) is a sensitive EGFR mutation or ALK fusion gene positive, required for first line progress after targeted therapy;Without mutations, required for first-line treatment;
4. Pemetrexed combined platinum did not progress by RECIST curative effect evaluation after 4 cycles of chemotherapy
5. ≥ 18 years of age ,Male or female
6. Eastern Cooperative Oncology Group(ECOG)performance scale 0 - 2.
7. Life expectancy of more than 3 weeks.
8. Adequate hepatic, renal, heart, and hematologic functions (Absolute Neutrophil Count(ANC) ≥ 1.5×109/L, Platelet (PLT) ≥ 100×109/L, Hemoglobin(HB) ≥ 100 g/L, total bilirubin within 1.5×the upper limit of normal(ULN), and serum transaminase≤2.5×the Upper Limit Of Normal(ULN), serum creatine ≤ 1 x Upper Limit Of Normal(ULN), creatinine clearance rate ≥ 50ml/min,
9. For women of child-bearing age, the pregnancy test results (serum or urine) within 7 days before enrolment must be negative. They will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men (previous surgical sterilization accepted), will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug.
10. Signed and dated informed consent. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

1. Squamous cell carcinoma (including adenosquamous carcinoma, undifferentiated carcinoma); small cell lung cancer (including small cell and non-small cell mixed lung cancer)
2. Genetic testing for sensitive EGFR mutation or ALK fusion gene is positive didn't accept targeted therapy
3. Symptomatic brain metastases (Patients who have no symptoms and is not needed to receive therapy before 21 days may participate in this trial, but need to be confirmed by MRI\CT or venography that no hematencephalon symptom);
4. Imaging (CT or MRI) shows that the tumor lesion vessels≤ 5 mm, or in the center of the large vessels tumor;Or show obvious lung empty or necrotic tumor;
5. Uncontrolled hypertension(systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mm Hg) even though two or more than two hypotensive agents application.
6. Patients who suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to New York Heart Association(NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%.
7. History of pulmonary interstitial diseases or concurrent pulmonary interstitial diseases.
8. Coagulation disfunction（INR>1.5 o rPT>Upper Limit Of Normal(ULN)+4s or Activated Partial Thromboplastin Time (APTT) >1.5 Upper Limit Of Normal(ULN)）, hemorrhagic tendency or receiving the therapy of thrombolysis or anticoagulation.
9. History of clinically significant haemoptysis =< 2 months (more than 2.5ml or half of one tea spoon of fresh blood per day) prior to registration.
10. History of clinically relevant major bleeding event=< 3 months.
11. Within 12 months before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack(TIA), hematencephalon, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.
12. Known inherited and acquired hemorrhagic and thromboplastic possibility (such as hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.)
13. Long-term untreated wounds or fractures.
14. Within 4 weeks of major surgery and/or injures, fractures , ulceration.
15. Significant factors that influence the ingestion and absorption of medicine, (e.g. unable swallow, chronic diarrhea and intestinal obstruction).
16. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess ≤ 6 months.
17. Urine protein≥++, or 24h urine protein quantitation≥1.0g.
18. History of psychiatric drugs abuse and not be abstinent, or dysphrenia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival（PFS） | Up to two years
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to two years

SECONDARY OUTCOMES:
Overall survival (OS) | Up to three years
  From date of randomization until the date of death from any cause, assessed up to three years
Objective response rate | Up to two years
  ORR is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments.
Disease control rate | Up to two years
  Investigators will assess treatment response according to Response Evaluation Criteria in Solid Tumors 1.1（RECIST1.1）
Adverse Events | Up to two years
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinqiao Hospital of Chongqing, Chongqing, China